CLINICAL TRIAL: NCT06712628
Title: Comparison of Persistence of UPadacitinib vs. TNF-inhibitoRs In a German Real-world SettING
Brief Title: A Comparison Study of Persistence of UPadacitinib vs. TNF-inhibitoRs In a German Real-world SettING
Acronym: UP-RISING
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-188
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Moderate to Severe Rheumatoid Arthritis
Keywords: Moderate to Severe Rheumatoid Arthritis; Rheumatoid Arthritis; Upadacitinib; Tumor Necrosis Factor Inhibitor Treatment
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Upadacitinib: Participants will receive upadacitinib as prescribed by their physician according to local label.
- Tumor Necrosis Factor Inhibitor-Treatment: Participants will receive a tumor necrosis factor inhibitor treatment as prescribed by their physician according to local label.

SUMMARY:
This study will compare the retention rates for UPA vs. TNFi treatment in adult participants with moderate to severe active RA per local label and according to local standard of care

This is a mono-country, prospective, multi-center observational study in patients with moderate to severe active RA receiving UPA or TNFi therapy. Around 678 participants will be enrolled in approximately 80 sites in Germany.

Study recruitment will last approximately 24 months, and the study participation time will be up to 24 months, for a total study duration of approximately 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Current or Past participants with a confirmed diagnosis of moderate to severe active RA upon judgement of the treating physician.
* Physician decision on participant treatment with Upadacitinib (UPA) or tumor necrosis factor inhibitor (TNFi) must have been reached prior to and independently of recruitment in the study
* UPA or TNFi prescribed in accordance with the applicable approved label and local regulatory and reimbursement policies

Exclusion Criteria:

* Participation in a clinical trial with an investigational drug (within a minimum of 30 days or 5 half-lives of the investigational drug [whichever is longer] prior to baseline)
* Prior treatment with Upadacitinib
* Prior treatment with the same tumor necrosis factor inhibitor as the one prescribed for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate to severe active Rheumatoid Arthritis receiving Upadcitinib or a Tumor necrosis factor inhibitor treatment.
Sampling Method: Non-Probability Sample
Enrollment: 678 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Retention Rate of UPA vs TNFi | Up to approximately 24 months
  Time to the discontinuation of Upadacitinib. Time to the discontinuation of Tumor Necrosis Factor Inhibitor treatment

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (52):
- Germany (52):
  - Gemeinschaftspraxis Innere Medizin/Rheumatologie /ID# 278584, Freiburg im Breisgau, Baden-Wurttemberg
  - Rheumapraxis Heidelberg /ID# 276475, Heidelberg, Baden-Wurttemberg
  - Rheumapraxis Haas Tübingen /ID# 275536, Tübingen, Baden-Wurttemberg
  - Rheumapraxis Ulm Dr. med. Nadia Rinaldi /ID# 276293, Ulm, Baden-Wurttemberg
  - Dr. Med. Thomas Marycz /ID# 274646, Amberg, Bavaria
  - Rheumapraxis Am Webereck /ID# 274412, Augsburg, Bavaria
  - Dr. Harmuth /ID# 273401, Marktredwitz, Bavaria
  - Praxiszentrum Dr. Med. Klaus Krüger Dres. Günther Kellerer Und Paul Kellerer /ID# 276138, Munich, Bavaria
  - Klinische Forschung Im Medizinischen Versorgungalltag Gbr /ID# 274587, Planegg, Bavaria
  - Private Practice - Dr. Dirk Wernicke /ID# 276820, Hohen Neuendorf, Brandenburg
  - Praxis K. Pagel /ID# 279121, Hoppegarten, Brandenburg
  - Rheumahaus Studien GbR /ID# 275917, Potsdam, Brandenburg
  - Rheumatologisch Immunologisch /ID# 275830, Templin, Brandenburg
  - Rheumatism Center Mittelhessen /ID# 274641, Bad Endenbach, Hesse
  - Deutsches Endokrinologisches Versorgungszentrum DEVZ - MVZ GdR /ID# 274291, Frankfurt am Main, Hesse
  - Rheumapraxis Hannover-List /ID# 273735, Hanover, Lower Saxony
  - Praxis. F. Bigdeli-Wilshusen /ID# 273455, Hanover, Lower Saxony
  - Rheumatologie Kassel /ID# 275916, Kassel, Lower Saxony
  - Rheumapraxis An Der Hase /ID# 276949, Osnabrück, Lower Saxony
  - Fachpraxis für Rheumatologie und Osteologie /ID# 275359, Weyhe, Lower Saxony
  - Private Practice - Dr. Thilo Klopsch - Stargarder Strasse /ID# 276367, Neubrandenburg, Mecklenburg-Vorpommern
  - Rheumazentrum Ruhrgebiet /ID# 275518, Herne, North Rhine-Westphalia
  - St.Elisabeth Hospital Meerbusch /ID# 275030, Meerbusch, North Rhine-Westphalia
  - Rheumazentrum Ratingen /ID# 275707, Ratingen, North Rhine-Westphalia
  - Praxis Dr. med. Florian Beyer /ID# 274293, Kaiserslautern, Rhineland-Palatinate
  - Rheumapraxis am Schlossberg /ID# 272728, Homburg, Saarland
  - Dr. Murawski /ID# 272724, Neunkirchen, Saarland
  - Knappschaftsklinikum Saar /ID# 279852, Püttlingen, Saarland
  - Rheumapraxis Dr. Prothmann /ID# 279851, Püttlingen, Saarland
  - Medizinischen Versorgungszentrums Agilomed /ID# 274887, Chemnitz, Saxony
  - Dr. Mueller /ID# 273081, Freiberg, Saxony
  - Private Practice - Dr. Frank Hamann, Dr. Andreas Teich & Dr. Konrad Boche /ID# 275358, Leipzig, Saxony
  - Private Practice - Dr. Ilka Schwarze /ID# 276981, Leipzig, Saxony
  - Private Practice - Dr. Christine Baumann /ID# 275095, Plauen, Saxony
  - Praxis H. Fricke-Wagner /ID# 274467, Zwickau, Saxony
  - Rheumapraxis Dr. Liebhaber /ID# 274888, Halle, Saxony-Anhalt
  - Rheumatologische Facharztpraxis /ID# 272866, Magdeburg, Saxony-Anhalt
  - Private Practice - Dr. Jochen Walter /ID# 280069, Rendsburg, Schleswig-Holstein
  - Private Practice - Dr. Thomas Kupka /ID# 273631, Altenburg, Thuringia
  - Rheumapraxis Weimar /ID# 272740, Weimar, Thuringia
  - MVZ Weserbergland /ID# 276009, Bad Pyrmont
  - Private Practice - Dr. Silke Zinke /ID# 276366, Berlin
  - MVZ Herzogin Elisabeth Hospital /ID# 272725, Braunschweig
  - Private Practice - Dr. Sebastian Schuh /ID# 272731, Coburg
  - Rheumapraxis Düren /ID# 272726, Düren
  - Praxis Dilltal /ID# 272727, Ehringshausen
  - Private Practice - Dr. Daniel Bestler /ID# 272741, Erfurt
  - Praxis Fiene /ID# 279410, Greifswald
  - Private Practice - Dr. Hauke E. Heintz /ID# 278081, Hamburg
  - Rheumatologische Facharztpraxis /ID# 272743, Naumburg
  - Cellitinnen-Krankenhaus St. Josef /ID# 275926, Wuppertal
  - Praxis Barmen /ID# 277514, Wuppertal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-188